CLINICAL TRIAL: NCT01666041
Title: Vascular and Metabolic Effects of Fenofibrate/Omega vs Fenofibrate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Kwang Kon Koh, professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMC-201202
Record Dates: First submitted 2012-08-15; First posted 2012-08-16 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2012-08

CONDITIONS: Hypertriglyceridemia
Keywords: insulin resistance
MeSH Terms: conditions — Hypertriglyceridemia; Insulin Resistance | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo
- fenofibrate/omega (Active Comparator): fenofibrate/omega
  Interventions: Drug: fenofibrate/omega
- fenofibrate (Active Comparator): fenofibrate
  Interventions: Drug: fenofibrate

INTERVENTIONS:
Drug: placebo
  Arms: placebo
Drug: fenofibrate/omega
  Arms: fenofibrate/omega
Drug: fenofibrate
  Arms: fenofibrate

SUMMARY:
The investigators hypothesize that fenofibrate/omega will improve insulin resistance compared with fenofibrate

ELIGIBILITY:
Inclusion Criteria:

* hypertriglyceridemia

Exclusion Criteria:

* moderate or severe hypertension, uncontrolled diabetes (HbA1c > 9%), nephrotic syndrome, hypothyroidism, coronary artery disease, or peripheral vascular disease

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
flow-mediated dilation | 8 weeks of treatment

SECONDARY OUTCOMES:
insulin resistance | 8 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Gil Medical Center, Incheon, South Korea